CLINICAL TRIAL: NCT04947995
Title: Validation of a Plasma-based Multiomics Assay and Risk Scoring Model for Screening of Gastric Malignancies
Brief Title: Multi-Omics Noninvasive Inspection of TumOr Risk for Gastric Cancer
Acronym: MONITOR- GAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GeneCast Biotechnology Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: D-P200110-MCCGW-HP-GC
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastric cancer group
  Interventions: Device: ctDNA multi-omics test
- Precancerous lesion group
  Interventions: Device: ctDNA multi-omics test
- Healthy group
  Interventions: Device: ctDNA multi-omics test

INTERVENTIONS:
Device: ctDNA multi-omics test — The ctDNA multi-omics test for gastric cancer will be built based on low-pass WGS, methylation, and target region sequencing.

SUMMARY:
This is a prospective, case-control study intended to develop and validate a blood-based multi-omics assay and computational model for early detection of gastric cancer. Approximately 450 subjects who receive esophageogastroscopy (EGD) will be enrolled and assigned to three arms including gastric cancer, precancerous lesion, and healthy control based on the diagnosis of EGD and histological results. Cell free DNA will be extracted from peripheral blood of all participants and assayed by next-generation sequencing for biomarkers including somatic mutation, methylation, and chromosome instability signals. In the first stage a multi-omics models will be developed for classification between malignancy group and control groups, and between precancerous group and healthy control. Sensitivity and specificity of the model will be evaluated in an independent validation group in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Age≥40
* Received EGD;
* Subjects must have given written informed consent, and the subjects compliance are good.

Exclusion Criteria:

* Subjects who could not accept EGD;
* Subjects who had previously undergone total or partial gastrectomy;
* There are other serious acute or chronic medical or mental diseases or laboratory abnormalities that may interfere with the interpretation of the research results and make the subjects unsuitable for the study in the judgment of the researchers;
* Subjects with a history of malignant tumor or two or more malignant tumors at the same time;
* Pregnant subjects;
* Subjects who had a history of bone marrow or organ transplantation, or had a history of blood transfusion one month before enrollment.
* The subjects with incomplete clinical data collection or other reasons judged by the researchers are not suitable for this study.

Ages: 40 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged≥40 who will receive EGD.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of blood-based multi-omics assay for early detection of gastric cancer with comparison to EGD and/or histological diagnosis. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No